CLINICAL TRIAL: NCT06558825
Title: Development and Pilot Testing of a Mental Health Clinic-Based PrEP Uptake and Adherence Intervention for Women in Treatment for Trauma-Related Conditions
Brief Title: Pre-exposure Prophylaxis (PrEP) Uptake and Adherence Intervention for Women with Trauma-related Conditions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Angela M Heads, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HSC-MS-21-0544; 1R34DA055496-01 (NIH)
Record Dates: First submitted 2024-08-14; First posted 2024-08-19 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Substance Use
Keywords: Pre-Exposure Prophylaxis; Women; HIV Prevention
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Integrated Intervention to Promote PrEP Uptake (Experimental)
  Interventions: Behavioral: Integrated Intervention to Promote PrEP Uptake
- Standard Treatment Condition (Active Comparator)
  Interventions: Other: Standard Treatment Condition

INTERVENTIONS:
Behavioral: Integrated Intervention to Promote PrEP Uptake — Provision of PrEP information through 3 counseling sessions, prevention navigation, and nurse practitioner-prescribed PrEP in an addiction treatment setting.
  Arms: Integrated Intervention to Promote PrEP Uptake
Other: Standard Treatment Condition — Participants in trauma treatment will be given information and referral to a community partner who will evaluate them to determine if they could benefit from PrEP for HIV prevention
  Arms: Standard Treatment Condition

SUMMARY:
The investigators have previously developed an integrated bio-behavioral intervention to promote PrEP uptake and adherence in cisgender women who are undergoing treatment for trauma-related mental health conditions and who are at a higher risk for HIV. The intervention is delivered within the mental health treatment setting and integrates knowledge, behavioral skills, and motivation to engage in and adhere to PrEP care. The purpose of this study is to assess the preliminary efficacy, feasibility, and acceptability of this intervention. The hypothesis is that, compared to standard treatment, the intervention will be feasible, acceptable, and associated with greater PrEP uptake and adherence.

ELIGIBILITY:
Inclusion Criteria:

* Currently undergoing mental health treatment;
* Have a history of trauma;
* HIV negative;
* Sexually active with an opposite sex partner within the past 6 months;
* Not using PrEP for HIV prevention at the time of screening;
* Eligible for PrEP based on having at least one Centers for Disease Control and Prevention (CDC)-defined criteria for PrEP;
* Fluent in English;
* Own or have regular access to a smart phone.

Exclusion Criteria:

* HIV positive;
* Concurrently participating in another HIV prevention program;
* Have severe cognitive impairment that would interfere with their ability to consent, understand study procedures and/or effectively participate in therapy;
* Have psychological distress that would prohibit them from participating in the study;
* Be unable or unwilling to meet study requirements.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants who uptake PrEP | 12 weeks post intervention
  PrEP uptake is defined as obtaining a prescription and taking the first dose.

SECONDARY OUTCOMES:
Number of Participants who adhere to PrEP | 12 weeks post PrEP initiation
  PrEP adherence is lab confirmed and is defined as having adequate levels of tenofovir (TFV) (>1000ng/ml).
PrEP adherence as assessed by proportion of videos uploaded | from the time of PrEP initiation to 12 weeks post PrEP initiation
  In the intervention arm, participants are asked to take a video of themselves taking PrEP. Videos are uploaded through an app, which is offered in the intervention arm only (and not the standard treatment arm). Data will be reported as the number of days a video is uploaded divided by the number of days of the intervention period.
PrEP adherence as assessed by proportion of self-reported daily adherence | from the time of PrEP initiation to 12 weeks post PrEP initiation
  In both arms, participants are sent a questionnaires weekly in which they record the number of days they took PrEP over the past seven days. Data will be reported as the number of days PrEP is taken divided by the number of days of the intervention period.
Intervention feasibility as assessed by number of participants enrolled | at the time of enrollment
  The number enrolled is the number of participants who signed the consent form.
Intervention feasibility as assessed by number of sessions attended by participants | 15 weeks post enrollment
Intervention feasibility as assessed by study retention | 15 weeks post enrollment
  Study retention is assessed by the the number of participants who completed the study.
Intervention acceptability as assessed by score on a satisfaction questionnaire | 15 weeks post enrollment
  This is a 15 item questionnaire and each item is scored from 1 (not at all true) to 9 (absolutely true). Total score ranges from 15 to 135, with a higher score indicating greater satisfaction.
Change in PrEP Anticipated Stigma as assessed by the PrEP Anticipated Stigma Scale | baseline, 15 weeks post enrollment
  Total score ranges from 8 to 32, with a higher score indicating greater stigma.
Change in perceived HIV risk as assessed by Perceived Risk of HIV Scale | baseline, 15 weeks post enrollment
  Total score ranges from 10 to 40, with a higher score indicating a greater perceived HIV risk.
Change in PrEP knowledge as assessed by PrEP Knowledge Questionnaire | baseline, 15 weeks post enrollment
  Total score ranges from 0 to 6, with a higher score indicating a greater knowledge about PrEP.
Change in PrEP attitudes as assessed by PrEP Attitudes Measure | baseline, 15 weeks post enrollment
  Total score ranges from 5.2 to 26, with a higher score indicating a better attitude toward PrEP.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Heads, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Louis A. Faillace, MD, Department of Psychiatry and Behavioral Sciences, University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No